CLINICAL TRIAL: NCT02024763
Title: Effect of an Educational Program on Schoolchildren's Energy Expenditure During Physical Education Classes
Brief Title: Educational Program and Schoolchildren's Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Paula Poblacion, Master in Science, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: APkit
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Physical Activity
Keywords: Energy Expenditure; Physical Education; Children; Randomized Controlled Trial
MeSH Terms: conditions — Motor Activity | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Intervention (Experimental): Intervention was applied to classroom teachers by the RRIDA Project team. Training lasted six weeks, 12 hours devoted to physical activity and 18 hours to nutritional content. Modules of educational activities were taught in order to be replicated at PE classes to 1st and 2nd grades' children of three exposed schools. Physical activity module was based on a theoretical approach of physical activity benefits and risks for health, children's physical fitness and activity patterns, physical education and change behavior models. In each meeting the PE professionals, performed PE classes with the classroom teachers as students, focusing in strategies to keep them in movement for the most of PE class time to stimulate students' joint participation instead of individual participation or games.
  Interventions: Behavioral: Educational Intervention
- No Intervention (No Intervention): No educational intervention was taken place in the control schools while the project was running. Afterwards, control schools received training.

INTERVENTIONS:
Behavioral: Educational Intervention — Intervention was applied to classroom teachers by the multidisciplinary team of the RRIDA Project. Training lasted six weeks, 12 hours devoted to physical activity and 18 hours to nutritional content. Modules of educational activities to classroom teachers were to be replicated at PE classes to children from 1st and 2nd grades of three exposed schools. The physical activity module was based on a theoretical approach of physical activity benefits and risks for health, children's physical fitness and activity patterns, physical education and change behavior models.
  Arms: Educational Intervention

SUMMARY:
The aim of this study was to evaluate the impact of a classroom teachers' educational intervention on 1st and 2nd grades children's physical activity level and energy expenditure during physical education classes in elementary public schools, in São Paulo, Brazil.

DETAILED DESCRIPTION:
This study is a School-based Randomized Controlled Trial. Three-step cluster sampling was used for subject selection. In the first step, 8 schools in the Vila Mariana district - São Paulo were selected and assigned randomly to physical activity intervention (3 schools) or control condition (5 schools). In the second step, all 48 classes from the 1st and 2nd grades were selected. In the third step, 352 children were randomly selected compose the observational group. In both groups, questionnaire data and SOFIT's observation were collected two times: "pre" (immediately before the intervention), and "post" (immediately after the intervention), with a six weeks interval between them. No educational intervention was taken place in the control schools while the project was running. Afterwards control schools received training.

ELIGIBILITY:
Inclusion Criteria:

* children from 7 to 10 years of age, enrolled at 1st or 2nd grades of selected schools in Vila Mariana - Sao Paulo.

Exclusion Criteria:

* Not have both observations.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 352 (Actual)
Dates: Start 1999-09; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Change in children's Physical Activity Level / Energy Expenditure after an Educational Intervention for classroom teachers. | Children's Physical Activity Level / Energy Expenditure were measured before and after an Educational Intervention to classroom teachers, with a six weeks interval.
  From eight elementary Public Schools we randomly selected three to receive an educational intervention for teachers. In order to evaluate intervention results, all the 1st and 2nd grades, from exposed and unexposed schools were nominated to have selected children. In each class, eight children were randomly selected. To assess children's level of physical activity, Physical Education classes were recorded. The videotapes analysis set the level of student's physical activity, teacher's attitude, and the class context. The observation instrument used was SOFIT - System for Observing Fitness Instruction Time. We analyzed and discussed the change in children's Physical Activity Level and Energy Expenditure before and after the Educational Intervention to classroom teachers, with a six weeks interval.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Augusto AC Taddei, MD, Dr PH, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil